CLINICAL TRIAL: NCT05020353
Title: A Study to Evaluate the Accuracy, Usability and Readability of the OraQuick® HIV Self-Test Performed by Observed Intended Users in Canada
Brief Title: OraQuick® HIV Self-Test Study in Canada
Acronym: OQHIVST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: REACH - HIV - OraQuick - 2.0
Record Dates: First submitted 2021-08-18; First posted 2021-08-25 (Actual); Results first posted 2025-05-11 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2024-05

CONDITIONS: HIV Testing; HIV Infections
Keywords: HIV; Self-testing; HIVST
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Intervention Model Description: Cross-sectional, prospective, field trial (untrained self-tester)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Investigational Device (Experimental): Observed self-test of oral fluid with the OraQuick HIV Self-Test
  Interventions: Device: OraQuick® HIV Self-Test

INTERVENTIONS:
Device: OraQuick® HIV Self-Test — OraQuick® HIV Self-Test in oral fluid conducted by observed intended users (non-healthcare professional and inexperienced in HIV self-testing) compared to laboratory 4th generation Ag/Ab enzyme immunoassay (EIA) results performed on venous blood.

SUMMARY:
Oral fluid based HIV Self-testing (HIVST) provides another innovative and simple option to increase opportunities for HIV testing. At-home testing for HIV using oral fluid has been FDA approved and in use in the USA since 2012, and studies have also shown that interest and acceptability of HIVST with oral fluid is high in other global settings. However data for oral fluid based HIVST within key populations and those at high risk for HIV infection in Canada is limited.

This study involves around 900 persons who are non-healthcare professionals and inexperienced in HIV self-testing (intended users) and are presenting at clinic sites across Canada for HIV testing. It will evaluate the accuracy (sensitivity and specificity), usability (persons performs test correctly) and readability (persons successfully interpret test results) of the OraQuick® HIV Self-Test when performed by persons representing intended users living in Canada.

A final report of study results will be provided to the Test manufacturer for inclusion in the Health Canada license application process.

DETAILED DESCRIPTION:
Background and Rationale:

Self-testing for HIV is an approach with the potential to increase the access, uptake and frequency of HIV testing for those who may not otherwise test and remain undiagnosed. There is increasing evidence showing the acceptability and usability of HIV self-testing (HIVST) in various key populations. In 2016 the World Health Organization recommended HIVST as an alternative option to complement existing HIV testing opportunities. Since then, HIVST use has been scaling up rapidly; for example, Canada's first blood-based (fingerstick) HIV self-test was licensed for use in November 2020.

Oral fluid based HIVST provides another innovative and simple option to increase opportunities for HIV testing. At-home testing for HIV using oral fluid has been FDA approved and in use in the USA since 2012, and studies have also shown that interest and acceptability of HIVST with oral fluid is high in other global settings. However data for oral fluid based HIVST within key populations and those at high risk for HIV infection in Canada is limited.

Having a licensed oral fluid HIV self-test in addition to the licensed blood-based HIV self-test will allow individuals to choose what is best for them and increase the potential to reach the undiagnosed living with HIV.

Objective:

This study will evaluate the accuracy, usability (persons performs test correctly) and readability (persons successfully interpret test results) of the OraQuick® HIV Self-Test when performed by persons representing intended users living in Canada.

Hypothesis:

The OraQuick Self-test as performed by intended users (non-healthcare professional and inexperienced in HIV self-testing) will meet or exceed the accuracy, usability and label comprehension requirements from Health Canada for license as a Class IV in vitro diagnostic device for Canadian market entry.

Study Design:

This study was designed around the requirements set out in the Health Canada Guidance Document: "Guidance for Manufacturers of Human Immunodeficiency Virus (HIV) Rapid Diagnostic Tests (RDT's) for Use at Point of Care or Self Testing, 2017". It is an investigational device trial designed as a cross-sectional study which employs observational and interview-based methods.

Sample population:

The study population requirements published by Health Canada stipulates that the prospective study include: 900 lay persons with unknown HIV status including 400 persons at risk for HIV infection (e.g. intravenous drug users, men who have sex with men, etc.). Self-reported practices or behaviour will be used to define those at high risk.

A minimum of 900 participants (non-healthcare professional and inexperienced in HIV self-testing) will read the instructions for use and conduct the OraQuick® HIV Self-Test. They will not be provided any training prior to use of the test. A trained healthcare provider or researcher (trained Observer) will watch, and document use of the test and independently read the participants self-test result. The participants will then complete a questionnaire to share their opinion on usability and label comprehension of this test.

A minimum of 400 (of the 900) participants will also be provided five mock devices with different results and asked to interpret those results i.e. strong positive; weak positive, negative, invalid with no control and no test line, and invalid with no control and a positive test line. This will evaluate readability of this test.

All participants will also have a venous blood sample collected for testing of plasma at a central laboratory with a 4th generation (Ag/Ab combo) HIV enzyme immunoassay that will serve as the comparator method (laboratory reference testing). All self-tests will be confirmed using a Canadian standard HIV testing algorithm. The sensitivity and specificity of the self-test result will be calculated relative to the "clinical truth" of the participants' HIV status determined by the confirmatory test process, where applicable. Participants will be instructed to return to the clinic for a follow-up visit, two (2) weeks after self-testing to obtain their laboratory test results which will be their official result.

Study Intervention Details:

Participants will be recruited to the study when they come in for voluntary HIV testing (e.g. POC testing) at a minimum of 3 study sites (different geographic locations). If persons consent to participating, all those enrolled will voluntarily complete a questionnaire (collecting demographics and HIV medical history information) and then provide their venous whole blood sample (for standard of care, laboratory confirmatory testing and comparator method), complete the OraQuick® HIV Self-Test (read test instructions, sample collection, sample testing, result interpretation), complete mock result interpretation, and complete questionnaires - Visit 1 (day 1; about 60 minutes). All patients will be instructed to return to the clinic for a follow-up visit two (2) weeks later to obtain their laboratory test results (Visit 2; about 15 - 60 minutes), post -test counselling, and to be linked to appropriate care depending on the test results..

Patients may also have a point-of-care (POC) test conducted on site as part of the clinic's standard of care testing, outside of the protocol and after all study procedures for Visit 1 are completed.

ELIGIBILITY:
Inclusion Criteria:

* Are 18 years of age and older
* Are able to speak / read / write English or French
* Have presented for voluntary testing for HIV infection in the clinic or community based setting
* Are willing to participate in the study site's standard of care HIV counselling and testing program and receive the study site's standard of care test results
* Are willing to be a participant in the study
* Are able to provide informed consent i.e. understands and signs the informed consent form
* Are able to complete the required testing on the allocated testing day
* Are willing to provide the necessary oral fluid and venipuncture blood for use in the study protocol testing methods.
* Are of unknown HIV status (last HIV negative test must be a minimum of 3 months prior)

Exclusion Criteria:

* Do not meet all the inclusion criteria
* Are known HIV positive
* Are on antiretroviral therapy (ART) or anti-HIV medications for the treatment of HIV, either as pre-exposure prophylaxis (PrEP), post-exposure prophylaxis (PEP) or experimental vaccine
* Have any experience or have ever conducted a rapid diagnostic self-test for HIV or any other sexually transmitted and blood borne illnesses disease
* Are currently participating in a concurrent trial of HIV self-tests
* Are investigator site employees or immediate family members of sponsor or investigator site employee
* Are a practicing medical healthcare professional (doctor, nurse or HIV counsellor that performs HIV testing with Rapid Tests)
* Any condition which, in the opinion of the Observer, would make the participant unsuitable or unsafe for enrolment or could interfere with the completion of the assessment and questionnaire etc. or bias the outcome, e.g. being unable to see / read by forgetting to bring reading glasses, being intoxicated, acute sickness, visibly distressed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 951 (Actual)
Dates: Start 2022-06-21 (Actual); Primary Completion 2023-07-04 (Actual); Study Completion 2024-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sean B Rourke, PhD, Principal Investigator — MAP Centre for Urban Health Solutions, St. Micheal's Hospital
Locations (7):
- Canada (7):
  - Cool Aid Community Health Centre, Vancouver, British Columbia
  - Nine Circles Community Health Centre, Winnipeg, Manitoba
  - ByWard Family Health Team, Ottawa, Ontario
  - Hassle Free Clinic, Toronto, Ontario
  - Maple Leaf Research, Toronto, Ontario
  - Women's Health in Women's Hands Community Health Centre, Toronto, Ontario
  - Clinique médicale l'Actuel, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Investigational Device
Started | 951
Completed | 911
Not Completed | 40
Not completed — Protocol Violation | 7
Not completed — Withdrawal by Subject | 33

BASELINE CHARACTERISTICS:
Population: Self-testing participants with unknown HIV status
Arm/Group | Investigational Device
Number analyzed (Participants) | 911
Age, Customized [Count of Participants; unit: Participants] — Population: Totals for each category varied based on participant responses
  Participants
    18-25 years | 307
    26-35 years | 302
    36-45 years | 158
    46-55 years | 73
    >55 years | 70
    Prefer not to answer | 1
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: Totals for each category varied based on participant responses
  Participants
    Cis-male | 434
    Cis-female | 450
    Other | 26
    Prefer not to anwer | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 911
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 235
  African/Caribbean/Black | 211
  Indigenous | 46
  Middle Eastern/North African | 25
  East Asian | 85
  South Asian | 222
  LatinX | 54
  Other | 33
Region of Enrollment [Count of Participants; unit: Participants]
  Canada: British Columbia | 102
  Canada: Manitoba | 56
  Canada: Ontario | 662
  Canada: Quebec | 91
Education [Count of Participants; unit: Participants] — Population: Totals for each category varied based on participant responses
  Participants
    No formal education | 0
    Primary school | 20
    Secondary school | 226
    College | 242
    University or higher | 420
    Prefer not to answer | 3
Employment [Count of Participants; unit: Participants] — Population: Totals for each category varied based on participant responses
  Participants
    Employed | 405
    Student | 261
    Retired | 23
    Unemployed | 215
    Prefer not to answer | 7
HIV Status [Count of Participants; unit: Participants]
  Negative status | 485
  Unknown status/never tested | 426
Medical Condition [Count of Participants; unit: Participants] — Population: Totals for each category varied based on participant responses
  Participants
    Diabetes | 21
    Hypertension | 23
    Sexually transmitted infection | 13
    Other medical condition | 86
    Answer not provided | 768
Reading/Writing Impairment [Count of Participants; unit: Participants] — Population: Totals for each category varied based on participant responses
  Participants
    No | 866
    Yes | 39
    Answer not provided | 6
Self-Reported HIV Risk [Count of Participants; unit: Participants]
  High risk | 520
  Low risk | 391
Sexual Orientation [Count of Participants; unit: Participants] — Population: Totals for each category varied based on participant responses
  Participants
    Heterosexual | 606
    Gay/Lesbian | 150
    Bisexual | 82
    Other | 52
    Prefer not to answer | 21
Tested for HIV Before [Count of Participants; unit: Participants] — Population: Totals for each category varied based on participant responses
  Participants
    No | 422
    Yes | 479
    Answer not provided | 10
Visual Impairment [Count of Participants; unit: Participants] — Population: Totals for each category varied based on participant responses
  Participants
    No | 604
    Yes | 301
    Answer not provided | 6

OUTCOME MEASURES:

1. Primary Outcome: Device Performance: Positive and Negative Percent Agreement
Description: Sensitivity and specificity of study participants' self-interpreted self-test results with the OraQuick® HIV Self-Test versus the HIV status as determined by the 4th generation EIA and confirmatory testing for HIV as necessary.
Time Frame: Outcome measured following POC tests on Visit 1, Day 1 for each participant.
Population: The invalids, inconclusive and not sure/do not know were not included in the calculations of Positive and Negative % Agreement.
Measure: Count of Participants; unit: Participants
Groups:
- Self-testing Participants: Unknown HIV status
Arm/Group | Self-testing Participants
Number analyzed (Participants) | 911
Participants
  True Positive | 1
  False Negative | 0
  True Negative | 880
  False Positive | 0
  Inconclusive | 1
  Positive % Agreement: number analyzed (Participants) | 1
  Positive % Agreement | 1
  Negative % Agreement: number analyzed (Participants) | 880
  Negative % Agreement | 880
  Invalid | 20
  Not sure/Do not know | 9

2. Primary Outcome: Observer Usability Assessment
Description: Observation to determine if participants perform all critical steps correctly
Time Frame: Outcome measured following POC tests on Visit 1, Day 1 for each participant.
Population: Totals for each category varied based on participant responses
Measure: Count of Units; unit: Expected Responses
Units Other Than Participants: Expected Responses
Arm/Group | Self-testing Participants
Number analyzed (Participants) | 906
Number analyzed (Expected Responses) | 906
Expected Responses
  Did the study participant read the instructions for use (IFU)?: Expected response | 859
  Did the study participant read the instructions for use (IFU)?: Unexpected response | 47
  Were the instructions for use (IFU) read before the test?: Expected response | 701
  Were the instructions for use (IFU) read before the test?: Unexpected response | 205
  Was the IFU referred to during the test process?: Expected response | 864
  Was the IFU referred to during the test process?: Unexpected response | 42
  Did the study participant remove the contents of the test pack?: Expected response | 901
  Did the study participant remove the contents of the test pack?: Unexpected response | 5
  Was the study participant able to find the test tube packet?: Expected response | 905
  Was the study participant able to find the test tube packet?: Unexpected response | 1
  Did the study participant remove the test tube from the packet?: Expected response | 905
  Did the study participant remove the test tube from the packet?: Unexpected response | 1
  Did the study participant remove the cap from the test tube?: Expected response | 896
  Did the study participant remove the cap from the test tube?: Unexpected response | 10
  Did the study participant place the test tube in the holder?: Expected response | 848
  Did the study participant place the test tube in the holder?: Unexpected response | 58
  Did the study participant have any difficulty with the test tube?: Expected response | 731
  Did the study participant have any difficulty with the test tube?: Unexpected response | 175
  Was the study participant able to find the test stick packet?: Expected response | 903
  Was the study participant able to find the test stick packet?: Unexpected response | 3
  Did the study participant remove the test stick from the packet?: Expected response | 902
  Did the study participant remove the test stick from the packet?: Unexpected response | 4
  Did the study participant touch the flat pad?: Expected response | 859
  Did the study participant touch the flat pad?: Unexpected response | 47
  Did the study participant collect the sample correctly (1x upper and lower swab)?: Expected response | 754
  Did the study participant collect the sample correctly (1x upper and lower swab)?: Unexpected response | 152
  Did the study participant place the test stick in the test tube correctly?: Expected response | 889
  Did the study participant place the test stick in the test tube correctly?: Unexpected response | 17
  Did the participant perform any steps out of the order?: Expected response | 800
  Did the participant perform any steps out of the order?: Unexpected response | 106
  Did the participant miss any step and continue the process despite a missed or incorrect step?: Expected response | 860
  Did the participant miss any step and continue the process despite a missed or incorrect step?: Unexpected response | 46
  Did the participant quit the process at any point?: Expected response | 905
  Did the participant quit the process at any point?: Unexpected response | 1
  Did the study participant wait 20 minutes before reading the results of the test?: Expected response | 820
  Did the study participant wait 20 minutes before reading the results of the test?: Unexpected response | 86

3. Primary Outcome: Participant and Observer Interpretations
Description: Confirmation by Observer to determine if participant interprets test results correctly and successful interpretation of various contrived (mock) test device results.
Time Frame: Outcome measured following POC tests on Visit 1, Day 1 for each participant.
Measure: Count of Participants; unit: Participants
Arm/Group | Self-testing Participants
Number analyzed (Participants) | 906
Participants
  Participant & Observer Agreement | 884
  Participant & Observer Disagreement | 22

4. Primary Outcome: Label Comprehension
Description: To determine that the participant is aware of key messages in labelling including test limitations and what to do following the test result.
Time Frame: Outcome measured following POC tests on Visit 1, Day 1 for each participant.
Population: The numbers are based on survey responses which varied across the different survey questions.
Measure: Count of Participants; unit: Participants
Arm/Group | Self-testing Participants
Number analyzed (Participants) | 911
Participants
  Did you use the Instructions for Use (IFU) sheet to help you complete the test?: number analyzed (Participants) | 903
  Did you use the Instructions for Use (IFU) sheet to help you complete the test?: Yes | 881
  Did you use the Instructions for Use (IFU) sheet to help you complete the test?: No | 22
  Were the Instructions for Use (IFU) easy to follow?: number analyzed (Participants) | 902
  Were the Instructions for Use (IFU) easy to follow?: Yes | 878
  Were the Instructions for Use (IFU) easy to follow?: No | 24
  Were the pictures and illustrations in the Instruction for Use (IFU) helpful?: number analyzed (Participants) | 902
  Were the pictures and illustrations in the Instruction for Use (IFU) helpful?: Yes | 878
  Were the pictures and illustrations in the Instruction for Use (IFU) helpful?: No | 24
  Was the Self-Test easy to use?: number analyzed (Participants) | 902
  Was the Self-Test easy to use?: Yes | 895
  Was the Self-Test easy to use?: No | 7
  Are you confident you could perform this test on your own?: number analyzed (Participants) | 902
  Are you confident you could perform this test on your own?: Yes | 899
  Are you confident you could perform this test on your own?: No | 3
  Would you use this test again if it were available to you?: number analyzed (Participants) | 902
  Would you use this test again if it were available to you?: Yes | 882
  Would you use this test again if it were available to you?: No | 20
  Would you prefer to use this test at home (yes) or get tested at a clinic (no)?: number analyzed (Participants) | 902
  Would you prefer to use this test at home (yes) or get tested at a clinic (no)?: Yes | 697
  Would you prefer to use this test at home (yes) or get tested at a clinic (no)?: No | 205
  Would you recommend this test to others? (e.g. a sexual partner, friend): number analyzed (Participants) | 902
  Would you recommend this test to others? (e.g. a sexual partner, friend): Yes | 890
  Would you recommend this test to others? (e.g. a sexual partner, friend): No | 12

5. Secondary Outcome: Readability or Interpretation (Mock Devices)
Description: The percentage of correct interpretations of contrived devices compared to the expected results.
Time Frame: Outcome measured following mock device interpretation on Visit 1, Day 1 for each participant.
Measure: Count of Units; unit: In Concordance
Units Other Than Participants: In Concordance
Arm/Group | Self-testing Participants
Number analyzed (Participants) | 465
Number analyzed (In Concordance) | 465
In Concordance
  Strong positive | 418
  Weak positive | 329
  Negative | 453
  Invalid, test line present | 273
  Invalid, no control line or test line | 448

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over the two week time frame in which the participant completed visit 1 and visit 2.
Arm/Group | Self-testing Participants
All-Cause Mortality (participants affected / at risk) | 0/951
Serious Adverse Events (participants affected / at risk) | 0/951
Other Adverse Events (participants affected / at risk) | 3/951
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Self-testing Participants (N=951)
Buffer solution-soaked swab placed in mouth (Product Issues) | 3 (3) — While conducting an HIV self-test in the OraQuick HIV Self-Test study, Participant placed the device swab into the test buffer solution before placing the buffer-soaked device into his/her mouth which is a procedure fault condition.

LIMITATIONS AND CAVEATS:
This is a prospective study for which the prevalence of infection is low.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-13): https://cdn.clinicaltrials.gov/large-docs/53/NCT05020353/Prot_SAP_000.pdf